CLINICAL TRIAL: NCT02889250
Title: Deep Brain Stimulation to Relieve Depression
Acronym: DRIVER
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: did not receive funding
Sponsor: Jordan F. Karp (Other)
Responsible Party: Sponsor-Investigator, Jordan F. Karp, Associate Professor of Psychiatry, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO16050040
Record Dates: First submitted 2016-08-13; First posted 2016-09-05 (Estimated); Last update posted 2018-08-06 (Actual); Status verified 2018-08

CONDITIONS: Treatment Resistant Depression
Keywords: geriatric; depression; deep brain stimulation; subcallosal cingulate
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Open Label DBS (Experimental): 6 months of DBS
  Interventions: Device: Medtronic Activa SC DBS, Lead Model 3387

INTERVENTIONS:
Device: Medtronic Activa SC DBS, Lead Model 3387 — Deep Brain Stimulation

SUMMARY:
This is an open label study with a sample size of 6 to develop deep brain stimulation of the subcallosal cingulate white matter(SCCWM) for late life depression using an experimental medicine approach in which the investigators will program the device based both on 1) a neurophysiologic measure of target engagement and 2) safety (defined as lack of neuropsychiatric worsening and stable neurocognition).

DETAILED DESCRIPTION:
Late-life treatment resistant depression (LL-TRD) is a public health and clinical dilemma.

Older patients with TRD are: 1) at greater risk for morbidity from medications and ECT, and 2) more likely to require maintenance ECT (which carries risks of cognitive impairment and repeated exposure to general anesthesia), compared to younger depressed patients. There is great need to develop targeted and safe treatments for those with LLTRD.

Deep brain stimulation (DBS) is a neurosurgical intervention with potential to become a treatment option for appropriately selected patients with LL-TRD. To date, the subcallosal cingulate white matter (SCCWM) is the DBS target with the most clinical, safety, and neurophysiologic data supporting therapeutic efficacy. The SCC is considered a "governor" for a network implicated in the processing of negative emotions and symptoms of depression. Furthermore, structural and functional impairments of the SCC and connected network structures are associated with LLD, supporting its potential as a target for DBS in older adults.

The overarching aim for this project is to develop DBS of the SCCWM for LL-TRD using an experimental medicine approach in which the investigators will program the device based both on 1) a neurophysiologic measure of target engagement and 2) safety (defined as lack of neuropsychiatric worsening and stable neurocognition). The proposed biomarker of target engagement is theta cordance (TC), a composite of absolute and relative theta power that is strongly correlated with regional neural metabolism. The hypothesis is that TC will increase during DBS is based on the observation of increased frontal TC during DBS in combination with PET data, which showed increased metabolism in frontal cortical structures in responders to DBS.

The investigators will use magnetoencephalography to measure TC during DBS and then will adjust stimulation settings to optimize target engagement over the course of the study, in response to observed increases in TC. Adding to the novelty of the project is use of personalized tractography to guide precise electrode placement in the area of the SCCWM which contain white matter tracts to mood-relevant frontal and subcortical nuclei.

During the two years of this open-label project the investigators will implant 6 patients. For each subject, over the course of 6 months, the investigators will ascertain the dose range effect of escalating DBS stimulation parameters on both TC and measures of safety.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed and dated the Screening Consent Form prior to conducting any study-related screening testing
2. Following successful completion of the screening phase, subject has signed and dated the Study Informed Consent Form prior to the initiation of any study-related procedures (other than screening testing).
3. Subject has been medically cleared for DBS neurosurgical procedure by their primary care doctor and study neurosurgeon.
4. Age >/= 60 years old.
5. Subject is fluent in English (written and verbal).
6. Subject meets Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for major depressive disorder (MDD) based on Structured Clinical Interview for DSM-5 Axis I Disorders (SCID-I) conducted during the screening testing for the project.
7. Subject has medical record documentation that the current major depressive episode (MDE) has persisted for > 2 years with the exception of brief responses (e.g., < 8 weeks) to treatments.
8. Subject's depression is treatment resistant; the subject has not clinical responded to 4 or more adequate drug trials of therapy for depression as scored by the antidepressant treatment history form.

   1. Three of the 4 trials need to have occurred in the current depressive episode.
   2. One of the 4 trials must have included a combination of 2 or more antidepressant medications from 2 different antidepressant classes.
   3. One of the 4 trials must have included 1 of the following: augmentation agents: lithium, triiodothyronine, buspirone, bupropion, or atypical antipsychotic.
9. Subject must have tried a course of ECT.
10. Subject's antidepressant medication regimen has been held stable for > 30 days prior to the study screening MADRS.
11. Subject's screening MADRS score > 25.
12. Average pre-operative MADRS score of 25 or greater (averaged over at least four weekly pre-surgical evaluations during the weeks prior to surgery) .
13. Aggregate score of > 8 on the social life and family life/home responsibilities subscales of the Sheehan Disability Scale.
14. Subject has received > 6 weeks of psychotherapy treatment, for the current or a previous depressive episode, without significant improvement.
15. Female subjects must not be pregnant, and if still of child bearing potential, must agree to a form of medically acceptable contraception.
16. If subject has a vagus nerve stimulator (VNS) implanted, they must agree to have the VNS system removed.
17. Subject agrees to not change psychotropic medication, psychotherapy, and outpatient psychiatric care program regimen throughout the screening phase and for the first six months after implantation of the DBS device.
18. Subject agrees to have the DRIVER investigators be the sole prescriber of psychotropic medications during the course of the study.
19. Evidence of connectivity (tractography identified streamlines) that is not disrupted by a significant burden of white matter hyperintensities between the SCC and nodes that may mediate response to DBS including MFC, dorsal and rostral cingulate, and subcortical nuclei.
20. Availability of an informant is required for study participation

Exclusion Criteria:

1. Inability to provide informed consent.
2. Inability to tolerate general anesthesia.
3. Subject has been hospitalized for treatment of depression < 30 days prior to the screening testing.
4. Active suicidal ideation with intent, suicide attempt within the last six months, or more than three suicide attempts within the last two years. Urgent psychiatric referral will be made in these cases.
5. Subject made a suicide attempt requiring medical treatment < 3 months prior to the screening testing.
6. Subject has a history of 2 or more suicide attempts < 12 months prior to the screening testing.
7. Subject poses an imminent suicide risk in the opinion of the investigator.
8. Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study that may confound the results of this study.
9. Subject has a history of a seizure disorder.
10. Subject will be exposed to diathermy.
11. Subject has a history of a neurosurgical ablation procedure.
12. Subject has a life expectancy of < 3 years.
13. Significant cerebrovascular risk factors or history of stroke, major head trauma, neurodegenerative disorder, or other general contraindications for DBS surgery (cardiac pacemaker/defibrillator or other Ferromagnetic implanted devices).
14. Contraindication to MRI.
15. Dementia, as defined by Modified Mini Mental State Examination (3MS) < 84 and clinical evidence of dementia. Patients screened out due to possible dementia will be referred to the local Memory Clinic or Alzheimer's Disease Research Center for evaluation to clarify the presence or absence of dementia.
16. Lifetime diagnosis of bipolar I or II disorder, schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, or current psychotic symptoms, obsessive compulsive disorder, panic disorder or post-traumatic stress disorder, or generalized anxiety disorder not secondary to the depression, as diagnosed by the SCID. A recommendation for psychiatric referral will be made in these cases.
17. Substance misuse (except for nicotine or caffeine) not in full sustained remission for at least one year as determined by SCID, and confirmed by study physician interview.
18. Anticoagulant pharmacotherapy.
19. Subjects that are determined during the screening phases to have severe personality disorders may be excluded.
20. Final patient selection will be made by consensus of the multidisciplinary study team. No exclusion criteria are based on race, ethnicity, or gender.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-06 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Theta cordance, measured by magnetoencephalography. | 6 months
  Theta cordance combines complementary information from absolute (the amount of power in the theta oscillatory band and relative power (the percentage of power contained in the theta band relative to the total spectrum) of EEG spectra.
Symptoms of Depression | 6 months
  A measure of safety is that the stimulation does not worsen depression. Significant worsening of depressive symptoms is defined as >/= 30% worsening of symptoms, as measured with the Montgomery Asberg Depression Rating Scale (MADRS) for four consecutive weeks, compared to the average score of the 4 weeks pre-stimulation.
Suicidality | 6 months
  A measure of safety is that the stimulation does not worsen or cause suicidal ideation or behavior. The Columbia Suicide Severity Rating Scale will assess suicidality. Clinically significant suicidality is defined as greater than 3 on suicidal ideation subscale of the Columbia Suicide Severity Scale AND worsening of the score compared to baseline, OR any suicidal behavior noted on the suicidal behavior subscale.
Neurocognitive status | 6 months
  A measure of safety is that the stimulation does not worsen neurocognition. The investigators will use a comprehensive validated battery of neuropsychiatric tests to monitor change in memory, executive functioning, psychomotor speed, verbal ability and global cognitive functioning. Clinically significant worsening is defined as deterioration of > 1 SD in at least two cognitive domains after six months of stimulation, compared to pre-surgical testing.

IPD SHARING:
Plan to Share IPD: Yes
The investigators will not share individual participant data. The investigators have a data sharing policy consistent with requirements of NIH.

REFERENCES:
- See also: Richardson RM, Ghuman AS, Karp JF. Results of the First Randomized Controlled Trial of Deep Brain Stimulation in Treatment-Resistant Depression. Neurosurgery. 2015 Aug;77(2):N23-4. — http://www.ncbi.nlm.nih.gov/pubmed/26181793
- See also: Alhourani A, McDowell MM, Randazzo MJ, Wozny TA, Kondylis ED, Lipski WJ, Beck S, Karp JF, Ghuman AS, Richardson RM. Network effects of deep brain stimulation. J Neurophysiol. 2015 Oct;114(4):2105-17. — http://www.ncbi.nlm.nih.gov/pubmed/26269552